CLINICAL TRIAL: NCT05778916
Title: Radiological Outcome vs.Patient Reported Clinical Outcome 5 Years Post Hallux Valgus Surgery
Brief Title: 5 Year Radiological and Clinical Results From Patients Operated for Hallux Valgus Deformity.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Ostfold Hospital Trust
Record Dates: First submitted 2022-11-28; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-11

CONDITIONS: Hallux Valgus
Keywords: Radiological outcome; Clinical outcome
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: 5 year follow up on patients operated for hallux valgus deformity — Clinical and radiological control of patients operated for hallux valgus deformity between 2016-2018.

SUMMARY:
Retrospective study of patients operated for hallux valgus deformity at our hospital (ostfold hospital trust) 5 years ago. Patients will be clinically examined, a weighted radiograph of the foot (traditional and newer parameters will be evaluated) and patient reported outcome measures (PROM) scores will be collected.

ELIGIBILITY:
Inclusion Criteria:

* All patients (18-80 years at time of surgery) operated for hallux valgus deformity at ostfold hospital trust 2016-2018

Exclusion Criteria:

* Not able to speak/write/read norwegian language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Norwegian speaking men and women operated for hallux valgus deformity at Ostfold hospital trust in the years 2016-2018.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-04-12 (Estimated); Primary Completion 2024-04-12 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical 5 year outcome | Data collection during 2023, completion during 2024
  Clinical (Manchester-oxford Foot Questionnaire (MOxFQ)

SECONDARY OUTCOMES:
Clinical VAS 5 year outcome | Data collection during 2023, completion during 2024
  Visual analogue scale (VAS 0-10)
Clinical Likert scale 5 year outcome | Data collection during 2023, completion during 2024
  Likert scale
Radiological outcomes | Until 2024
  Measurement of correction

CONTACTS AND LOCATIONS:
Overall Officials: Marius Molund, MD, phd, Study Director — Ostfold Hospital Trust
Locations (1):
- Østfold Hospital Trust, Sarpsborg, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: Undecided